CLINICAL TRIAL: NCT06784804
Title: Objective vs. Subjective Physical Activity Assessment in a Clinical Setting of Patients With Obesity and Comorbid Eating Disorders
Brief Title: Comparing Objective and Subjective Physical Activity Assessments in Obese Patients
Acronym: OSPAA
Status: Completed | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Patrick Kutschar, Ass. Prof. Mag. Dr. Patrick Kutschar, Paracelsus Medical University
Other Study IDs: OSPAA-Obesity
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Physical Activity; Anorexia Nervosa; Bulimia Nervosa; Obesity
Keywords: Concurrent validity; SenseWear Actigraph; IPAQ-SF; Exercise therapy; Obesity; Self-report bias
MeSH Terms: conditions — Motor Activity; Anorexia Nervosa; Bulimia Nervosa; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Obese patients with anorexia nervosa or bulimia nervosa: Patients admitted during the study period were eligible if they were ≥ 18 years old, had a body mass index (BMI) ≥ 30, could read and speak German, had a diagnosis of an eating disorder (ICD-10: F50.9 unspecified eating disorder, F50.2 bulimia nervosa), had a clinical stay of at least 4 weeks, and wore the SWA for at least 18 h·d-1, including at least 4 days with one weekend day.
  Participant characteristics were as follows:
  Sex (f/m) 23 (17/6) Age (f/m) 42.1 ± 13.6 BMI (kg·m-2) 40,5 ± 5.7 Body fat (%) 43.5 ± 6.8 Sleep efficiency 81 ± 8 SWA wearing time 1400 ± 43 Activity in min (>3 MET) 94 ± 37 Steps 9935 ± 3050 Clinical stay (d) 61 ± 16 Eating disorders Eating disorder, F50.9 (%) 91 Bulimia nervosa, F50.2 (%) 9 Psychosomatic disorders Depression, F33 (%) 26 Personality disorders, F60 (%) 17 Neurotic disorders, F4 (%) 30 Bipolar disorders F31 (%) 4

SUMMARY:
The goal of this observational study is to analyze the validity of self-reported physical activities in obese patients with psychosomatic disorders in a clinical setting. The main question aims to answer:

- How valid are self-reported physical activity data (via the International Physical Activity Questionnaire, IPAQ-SF) compared to actigraphy-based objective measurements (using the SenseWear® armband, SWA)?

Between 2020 and 2022, 23 patients with obesity (21 anorexia nervosa, 2 bulimia nervosa) were recruited from an Austrian psychosomatic clinic. Receiving routine care, participants were additionally asked to

* wear the SWA for seven days in the clinic
* complete the IPAQ-SF for the same reference period on the first weekday after SWA wearing time

The study then statistically compared total physical activity, measured in so called metabolic equivalents (MET minutes per week), and sitting time (minutes per day) between the two methods to determine the accuracy of the self-reported data.

DETAILED DESCRIPTION:
This methodological study presents the effort of a collaboration between the Department of Sport and Exercise Science (Paris Lodron University, Salzburg), the Psychosomatic Clinic Eggenburg (Eggenburg, Lower Austria, Austria), and the Paracelsus Medical University (Salzburg, Austria). The empirical work was done by a Master Student as part of a scientific qualification work (M.A. Sports Physiotherapy MSc) and supervised by a member of the research team.

Rationale of the Study:

Accurate measurement of physical activity is essential for addressing obesity, treating eating disorders, and combating the broader obesity epidemic. However, effective treatment requires accurate activity assessments. Traditional self-reported questionnaires often fail to provide this accuracy, particularly in populations where physical or psychological factors impair recall accuracy.

For patients treated for obesity and psychosomatic eating disorders, recall impairments are likely further exacerbated by distorted perceptions of normal physical activity, as well as stress, shame, stigmatization, and guilt.

Moreover, we expect the extent of inaccuracy in self-reported activity duration, frequency or intensity to depend on the actual magnitude of activity.

No previous study has focused on this population or used concurrent validity analysis to compare subjective vs objective measures of physical activity while addressing potential proportional bias adequately.

Hence, valid measurement of physical activity is crucial for treating obesity, eating disorders, and combating the obesity epidemic.

In this methodological study, the investigators assess the concurrent validity of self-reported questionnaires and actigraph-based objective measurements of physical activity in patients with obesity and psychosomatic eating disorders in a clinical setting. As a secondary aim, this research will evaluate potential moderator effects of obesity level and sex. Given its role as an objective measure, the sensor-based actigraph was used as a criterion to validate the IPAQ. The investigators hypothesize that subjective self-reports from the IPAQ will overestimate total physical activity, but underestimate sitting time compared to objective actigraph data.

Applied methods:

A concurrent validity study was conducted at the Psychosomatic Clinic in Eggenburg (Austria) from May 2020 to March 2022. In total, 23 obese patients (17 female, 6 male; 42 ± 14 years; BMI 41 ± 6 kg·m-2, 21 diagnosed with anorexia nervosa (ICD-10: F50.9), 2 with bulimia nervosa (ICD-10: F50.2), were recruited from an Austrian psychosomatic clinic. Patients admitted during the study period were eligible if they were ≥ 18 years old, had a body mass index (BMI) ≥ 30, could read and speak German, had a diagnosis of an eating disorder (ICD-10: F50.9 unspecified eating disorder, F50.2 bulimia nervosa), had a clinical stay of at least 4 weeks, and wore the SWA for at least 18 h·d-1, (41) including at least 4 days with one weekend day.

Patients self-administered the International Physical Activity Questionnaire (IPAQ-SF) while wearing the SenseWear® armband (SWA) for 7 days during the 3rd to 4th week of their clinical stay. Outcome measures included total physical activity, assessed using metabolic equivalents (MET min·w-1) and sitting time (min·d-1).

Concurrent validity - SWA as a criterion - was assessed using regression analyses, and proportional bias was examined through regression and equality line similarity analyses.

Expected benefits:

Valid information about physical activity is key for treating adults with obesity and psychosomatic disorders. The study will add further evidence to the of validity of self-reported physical activity. For the first time, concurrent validity of the specific population of obese patients is studied. The study results will help to better and more precise measure and estimate physical activity in obese patients. This will be crucial to informing intervention and treatment programs in practice as well as shed further light on how to measure the patient reported activity level in the most accurate and valid way.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* body mass index (BMI) ≥ 30
* could read and speak German
* had a diagnosis of an eating disorder (ICD-10: F50.9 unspecified eating disorder, F50.2 bulimia nervosa)
* had a clinical stay of at least 4 weeks
* wore the SWA for at least 18 h·d-1, (41) including at least 4 days with one weekend day

Exclusion Criteria:

* inability to walk independently
* a nickel allergy
* valid wearing time of accelerometer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 23 patients at the Psychosomatic Clinic in Eggenburg (Austria) from May 2020 to March 2022 were recruited.
  Patients received standardized instructions about the study's purpose and the use of the SWA and IPAQ-SF. During the first two weeks, they followed standard clinic therapies, including exercise. Body fat was measured before activity monitoring began. The SWA was provided during week three or four, with instructions on use and activity logging. Patients also completed the IPAQ-SF for the prior week. They were advised to maintain normal activity patterns and record non-wearing periods. Blinding was not feasible.
  Patients provided written informed consent to participate and for the use of their data in research. The patients were informed in detail about the study procedures. Participants took part in the study voluntarily and had the option of withdrawing at any time. Their privacy and rights were carefully protected throughout the study..
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
MET (Metabolic equivalents) - Objective measure of physical activity in MET min/week (by SWA) | Period: SWA was worn for at least four days within week 3 or week 4 of clinical stay
  The lightweight (83 g) SenseWear® Armband Pro 3 (Bodymedia, Inc., Pittsburgh, PA, USA) is a multisensory device that includes a two-axis accelerometer, as well as sensors to measure galvanic skin responses, skin and ambient temperature or heat flux. The monitor was initialized based patient's gender, age, weight and height, and was adjusted to fit on the triceps muscle, halfway between the acromion and olecranon processes of the dominant arm. A proprietary algorithm converts raw data into estimates of total and active energy expenditure, resting metabolic rate, metabolic units, total number of steps, duration of physical activity, duration of sleep and resting time. Data are expressed both in kcal·min-1 and metabolic equivalents (METs). The time of physical activity is categorized into different ranges based on the metabolic equivalent (MET). Values <3 MET are classified as low, METs between 3 and 6 as moderate values ≥6 MET as vigorous activity.
MET (Metabolic equivalent) - Subjective measure of physical activity in MET min/week (by IPAQ self-report) | Single time point: Retrospective self-report on the first weekday after SWA wearing time
  The International Physical Activity Questionnaire Short Form (IPAQ-SF) provides a standardized measure of physical activity for individuals across different populations. The most used short form consists of seven items that assess physical activity (frequency, duration) over the past seven days, categorizing it into four types: vigorous intensity, moderate intensity, walking, and sitting. An average metabolic equivalents score (MET, min·w-1) was calculated to assess total physical activity as well as for each type of activity, separately. For walking activities, all types of walking were included and an average MET score was derived. The same procedure was carried out for medium intensity and high intensity activities. By calculating the number of activity days multiplied by the average duration per activity, statements about the energy consumption per week and the fitness level can be derived. The last seven days in which the SWA was worn were used as the reference period.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Wiesinger, PhD, Principal Investigator — Paracelsus Medical University; Elmar Kaiser, Dr. med., Chief physician, Principal Investigator — Psychosomatic Clinic Eggenburg; Bettina Bannert, MA, Principal Investigator — Psychosomatic Clinic Eggenburg
Locations (1):
- Psychosomatic Clinic Eggenburg, Eggenburg, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided